CLINICAL TRIAL: NCT02425644
Title: Multicenter, Randomized, Double-blind, Parallel-group, Active-controlled, Superiority Study to Compare the Efficacy and Safety of Ponesimod to Teriflunomide in Subjects With Relapsing Multiple Sclerosis
Brief Title: Oral Ponesimod Versus Teriflunomide In Relapsing MUltiple Sclerosis
Acronym: OPTIMUM
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Actelion (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AC-058B301; 2012-000540-10 (EudraCT Number)
Record Dates: First submitted 2015-04-21; First posted 2015-04-24 (Estimated); Results first posted 2021-06-11 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Multiple Sclerosis
Keywords: relapsing multiple sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — ponesimod; teriflunomide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Ponesimod (Experimental): Subjects to receive 20 mg ponesimod
  Interventions: Drug: ponesimod
- Teriflunomide (Active Comparator): Subjects to receive 14 mg teriflunomide
  Interventions: Drug: teriflunomide

INTERVENTIONS:
Drug: ponesimod — film-coated tablet with 20 mg ponesimod, administered orally once daily in the morning
  Other Names: ACT-128800
  Arms: Ponesimod
Drug: teriflunomide — film-coated tablet with 14 mg teriflunomide, administered orally once daily in the morning
  Arms: Teriflunomide

SUMMARY:
International clinical trial to compare ponesimod and teriflunomide in relapsing multiple sclerosis

ELIGIBILITY:
Inclusion Criteria:

Male and female subjects aged 18 to 55 years with established diagnosis of MS McDonald 2010 with relapsing course from onset (i.e., RRMS and SPMS with superimposed relapses).

Subjects must have active disease evidenced by one or more MS attacks with onset within the period of 12 to 1 months prior to randomization, or by two or more MS attacks with onset within the 24 to 1 months prior to randomization, or with one or more gadolinium-enhancing (Gd+) lesion(s) of the brain on an MRI performed within 6 months prior to randomization.

Enrolled subjects must be ambulatory (EDSS score of up to 5.5 inclusive) and may be treatment-naïve or previously treated with MS disease modifying therapy.

Exclusion Criteria:

Subjects with significant medical conditions or therapies for such conditions (e.g., cardiovascular, pulmonary, immunological, hepatic,ophthalmological conditions) or lactating or pregnant women are not eligible to enter the study.

Subjects with contraindications to MRI or with clinically relevant medical or surgical conditions that, in the opinion of the investigator, would put the subject at risk by participating in the study are not eligible to enter the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1133 (Actual)
Dates: Start 2015-06-04 (Actual); Primary Completion 2019-05-16 (Actual); Study Completion 2019-05-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tatiana Scherz, MD, PhD, Study Director — Actelion
Locations (162):
- United States (10):
  - Investigator Site 8045, Carlsbad, California
  - Investigator Site 8311, Pomona, California
  - Investigator Site 8036, Denver, Colorado
  - Investigator Site 8065, Ormond Beach, Florida
  - Investigator Site 8018, Tampa, Florida
  - Investigator Site 8013, Indianapolis, Indiana
  - Investigator Site 8040, Raleigh, North Carolina
  - Investigator Site 8006, Columbus, Ohio
  - Investigator Site 8015, Franklin, Tennessee
  - Investigator Site 8042, Orem, Utah
- Belarus (5):
  - Investigator Site 3605, Grodno
  - Investigator Site 3603, Minsk
  - Investigator Site 3602, Minsk
  - Investigator Site 3606, Vitebsk
  - Investigator Site 3604, Vitebsk
- Investigator Site 9104, Sarajevo, Bosnia and Herzegovina
- Bulgaria (7):
  - Investigator Site 2709, Plovdiv
  - Investigator Site 2711, Sofia
  - Investigator Site 2702, Sofia
  - Investigator Site 2707, Sofia
  - Investigator Site 2701, Sofia
  - Investigator Site 2708, Sofia
  - Investigator Site 2703, Sofia
- Canada (4):
  - Investigator Site 8102, Edmonton, Alberta
  - Investigator Site 8120, Victoria, British Columbia
  - Investigator Site 8101, Ottawa, Ontario
  - Investigator Site 8113, Greenfield Park, Quebec
- Croatia (4):
  - Investigator Site 2506, Osijek
  - Investigator Site 2502, Zagreb
  - Investigator Site 2508, Zagreb
  - Investigator Site 2509, Zagreb
- Czechia (9):
  - Investigator Site 3009, Brno
  - Investigator Site 3003, Brno
  - Investigator Site 3010, Hradec Králové
  - Investigator Site 3006, Jihlava
  - Investigator Site 3002, Ostrava-Poruba
  - Investigator Site 3007, Pardubice
  - Investigator Site 3001, Prague
  - Investigator Site 3008, Prague
  - Investigator Site 3004, Teplice
- Finland (2):
  - Investigator Site 2212, Tampere
  - Investigator Site 2202, Turku
- France (5):
  - Investigator Site 1713, Bordeaux
  - Investigator Site 1703, Clermont-Ferrand
  - Investigator Site 1715, Nantes
  - Investigator Site 1706, Nice
  - Investigator Site 1705, Strasbourg
- Georgia (5):
  - Investigator Site 3905, Tbilisi
  - Investigator Site 3904, Tbilisi
  - Investigator Site 3903, Tbilisi
  - Investigator Site 3906, Tbilisi
  - Investigator Site 3902, Tbilisi
- Germany (5):
  - Investigator Site 1113, Dresden
  - Investigator Site 1107, Erfurt
  - Investigator Site 1109, Leipzig
  - Investigator Site 1104, Mainz
  - Investigator Site 1102, Ulm
- Greece (3):
  - Investigator Site 1303, Athens
  - Investigator Site 1301, Athens
  - Investigator Site 1307, Athens
- Hungary (5):
  - Investigator Site 2903, Budapest
  - Investigator Site 2905, Budapest
  - Investigator Site 2910, Esztergom
  - Investigator Site 2902, Győr
  - Investigator Site 2909, Kistarcsa
- Israel (4):
  - Investigator Site 4005, Ashkelon
  - Investigator Site 4004, Haifa
  - Investigator Site 4006, Jerusalem
  - Investigator Site 4010, Zfat
- Italy (4):
  - Investigator Site 1403, Cefalù
  - Investigator Site 1409, Genova
  - Investigator Site 1413, L’Aquila
  - Investigator Site 1405, Roma
- Latvia (3):
  - Investigator Site 3401, Riga
  - Investigator Site 3402, Riga
  - Investigator Site 3403, Riga
- Lithuania (3):
  - Investigator Site 3502, Kaunas
  - Investigator Site 3503, Klaipėda
  - Investigator Site 3504, Šiauliai
- Mexico (2):
  - Investigator Site 7410, Chihuahua City
  - Investigator Site 7409, Monterrey
- Poland (12):
  - Investigator Site 3219, Bialystok
  - Investigator Site 3215, Bydgoszcz
  - Investigator Site 3208, Gdansk
  - Investigator Site 3217, Katowice
  - Investigator Site 3203, Katowice
  - Investigator Site 3205, Konstancin-Jeziorna
  - Investigator Site 3216, Ksawerów
  - Investigator Site 3220, Lublin
  - Investigator Site 3202, Poznan
  - Investigator Site 3214, Poznan
  - Investigator Site 3207, Poznan
  - Investigator Site 3213, Wroclaw
- Portugal (4):
  - Investigator Site 1602, Amadora
  - Investigator Site 1605, Braga
  - Investigator Site 1603, Coimbra
  - Investigator Site 1604, Porto
- Romania (4):
  - Investigator Site 2807, Bucharest
  - Investigator Site 2811, Bucharest
  - Investigator Site 2804, Bucharest
  - Investigator Site 2802, Timișoara
- Russia (28):
  - Investigator Site 3821, Barnaul, Altayskiy Kray
  - Investigator Site 3818, Belgorod
  - Investigator Site 3837, Bryansk
  - Investigator Site 3811, Kazan'
  - Investigator Site 3822, Kemerovo
  - Investigator Site 3814, Krasnoyarsk
  - Investigator Site 3823, Kursk
  - Investigator Site 3831, Moscow
  - Investigator Site 3803, Moscow
  - Investigator Site 3840, Moscow
  - Investigator Site 3810, Moscow
  - Investigator Site 3834, Nizhny Novgorod
  - Investigator Site 3802, Nizhny Novgorod
  - Investigator Site 3829, Novosibirsk
  - Investigator Site 3839, Perm
  - Investigator Site 3812, Pyatigorsk
  - Investigator Site 3808, Saint Petersburg
  - Investigator Site 3833, Saint Petersburg
  - Investigator Site 3813, Saint Petersburg
  - Investigator Site 3807, Saint Petersburg
  - Investigator Site 3815, Saint Petersburg
  - Investigator Site 3805, Samara
  - Investigator Site 3825, Smolensk
  - Investigator Site 3801, Tomsk
  - Investigator Site 3819, Tver'
  - Investigator Site 3835, Veliky Novgorod
  - Investigator Site 3842, Yaroslavl
  - Investigator Site 3836, Yekaterinburg
- Serbia (5):
  - Investigator Site 2601, Belgrade
  - Investigator Site 2606, Belgrade
  - Investigator Site 2607, Belgrade
  - Investigator Site 2603, Kragujevac
  - Investigator Site 2602, Niš
- Spain (6):
  - Investigator Site 1509, Barcelona
  - Investigator Site 1505, Barcelona
  - Investigator Site 1504, Barcelona
  - Investigator Site 1502, Madrid
  - Investigator Site 1501, Málaga
  - Investigator Site 1506, Seville
- Sweden (3):
  - Investigator Site 2103, Gothenburg
  - Investigator Site 2110, Stockholm
  - Investigator Site 2101, Stockholm
- Investigator Site 9004, Trabzon, Turkey (Türkiye)
- Ukraine (15):
  - Investigator Site 3714, Chernihiv
  - Investigator Site 3701, Chernihiv
  - Investigator Site 3713, Ivano-Frankivsk
  - Investigator Site 3711, Ivano-Frankivsk
  - Investigator Site 3723, Kharkiv
  - Investigator Site 3724, Kharkiv
  - Investigator Site 3716, Kyiv
  - Investigator Site 3715, Lviv
  - Investigator Site 3721, Lviv
  - Investigator Site 3703, Odesa
  - Investigator Site 3717, Poltava
  - Investigator Site 3730, Ternopil
  - Investigator Site 3718, Vinnytsia
  - Investigator Site 3722, Zaporizhia
  - Investigator Site 3725, Zhytomyr
- United Kingdom (3):
  - Investigator Site 2015, Glasgow
  - Investigator Site 2021, Lancashire
  - Investigator Site 2003, Salford

REFERENCES:
- [Derived] Jones RR, Turkoz I, Ait-Tihyaty M, DiBernardo A, Houtchens MK, Havrdova EK. Efficacy and Safety of Ponesimod Compared with Teriflunomide in Female Patients with Relapsing Multiple Sclerosis: Findings from the Pivotal OPTIMUM Study. J Womens Health (Larchmt). 2024 Apr;33(4):480-490. doi: 10.1089/jwh.2023.0037. Epub 2024 Feb 1. PMID 38301149
- [Derived] Jiang T, Ziemssen T, Wray S, Shen C, Soderbarg K, Lewin JB, Bozin I, Freedman MS. Matching-Adjusted Indirect Comparisons of Diroximel Fumarate, Ponesimod, and Teriflunomide for Relapsing Multiple Sclerosis. CNS Drugs. 2023 May;37(5):441-452. doi: 10.1007/s40263-023-01002-x. Epub 2023 May 8. PMID 37155132
- [Derived] Fox RJ, Tervonen T, Phillips-Beyer A, Sidorenko T, Boyanova N, Brooks A, Hennessy B, Jamieson C, Levitan B. The relevance of fatigue to relapse rate in multiple sclerosis: Applying patient preference data to the OPTIMUM trial. Mult Scler. 2023 Mar;29(3):427-435. doi: 10.1177/13524585221140270. Epub 2022 Dec 22. PMID 36550636
- [Derived] Valenzuela B, Olsson Gisleskog P, Poggesi I, Sidorenko T, Burcklen M, Kracker H, Perez-Ruixo JJ. An exposure-response analysis of ponesimod clinical efficacy in a randomized phase III study in patients with relapsing multiple sclerosis. CPT Pharmacometrics Syst Pharmacol. 2022 Oct;11(10):1294-1304. doi: 10.1002/psp4.12778. Epub 2022 Sep 1. PMID 36047474
- [Derived] Kappos L, Fox RJ, Burcklen M, Freedman MS, Havrdova EK, Hennessy B, Hohlfeld R, Lublin F, Montalban X, Pozzilli C, Scherz T, D'Ambrosio D, Linscheid P, Vaclavkova A, Pirozek-Lawniczek M, Kracker H, Sprenger T. Ponesimod Compared With Teriflunomide in Patients With Relapsing Multiple Sclerosis in the Active-Comparator Phase 3 OPTIMUM Study: A Randomized Clinical Trial. JAMA Neurol. 2021 May 1;78(5):558-567. doi: 10.1001/jamaneurol.2021.0405. PMID 33779698
- See also: Multicenter, randomized, double-blind, parallel-group, active-controlled, superiority study to compare the efficacy and safety of ponesimod to teriflunomide in subjects with relapsing multiple sclerosis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217051&parentIdentifier=AC-058B301&attachmentIdentifier=24f4f084-9a98-4430-a172-80d455f49865&fileName=AC-058B301_Additional_result_data_CH.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: As planned, Placebo was not a separate arm as this was included for double dummy design study part (up to Day 14).
Groups:
- Ponesimod 20 mg: Participants were up-titrated during Days 1 to 14 from 2 to 10 mg of ponesimod once daily (one ponesimod tablet and one matching placebo capsule per day). From Day 15 to Week 108 participants received ponesimod 20 mg once daily up to Week 108
- Teriflunomide 14 mg: Participants received teriflunomide 14 mg capsule once daily from Day 1 up to Week 108. During Days 1 to 14 (mock uptitration period), participants received in addition one tablet of matching placebo.
Period: Overall Study
Arm/Group | Ponesimod 20 mg | Teriflunomide 14 mg
Started | 567 | 566
Treated | 565 | 566
Completed | 490 | 495
Not Completed | 77 | 71
Not completed — Lost to Follow-up | 2 | 3
Not completed — Withdrawal by Subject | 41 | 36
Not completed — Lack of Efficacy | 3 | 10
Not completed — Adverse Event | 13 | 3
Not completed — Death | 0 | 2
Not completed — Other | 18 | 17

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ponesimod 20 mg | Teriflunomide 14 mg | Total
Number analyzed (Participants) | 567 | 566 | 1133
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.7 (8.74) | 36.8 (8.74) | 36.7 (8.74)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 363 | 372 | 735
  Male | 204 | 194 | 398
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 2 | 5
  White | 551 | 553 | 1104
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 13 | 10 | 23
Region of Enrollment [Count of Participants; unit: Participants]
  BELARUS | 21 | 24 | 45
  BULGARIA | 18 | 27 | 45
  CANADA | 10 | 7 | 17
  CROATIA | 14 | 20 | 34
  CZECH REPUBLIC | 55 | 46 | 101
  FINLAND | 4 | 3 | 7
  FRANCE | 8 | 8 | 16
  GEORGIA | 24 | 17 | 41
  GERMANY | 9 | 7 | 16
  GREECE | 9 | 6 | 15
  HUNGARY | 7 | 12 | 19
  ISRAEL | 4 | 9 | 13
  ITALY | 7 | 7 | 14
  LATVIA | 11 | 4 | 15
  LITHUANIA | 3 | 8 | 11
  MEXICO | 7 | 10 | 17
  POLAND | 80 | 71 | 151
  PORTUGAL | 10 | 10 | 20
  ROMANIA | 10 | 5 | 15
  RUSSIAN FEDERATION | 116 | 111 | 227
  SPAIN | 34 | 39 | 73
  SWEDEN | 8 | 6 | 14
  TURKEY | 2 | 0 | 2
  UKRAINE | 57 | 66 | 123
  UNITED KINGDOM | 2 | 5 | 7
  UNITED STATES | 22 | 17 | 39
  Serbia | 14 | 19 | 33
  Bosnia | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Annualized Confirmed Relapse Rate
Description: Relapse: occurrence of acute episode of one or more new symptoms or worsened symptoms of Multiple sclerosis (MS), not associated with fever/infection and lasting 24 hours after stable 30 days period. Confirmed relapse: increase from baseline at least 0.5 point Expanded Disability Status Scale (EDSS) score or increase of one point in one, two or three Functional Systems (FS), excluding bowel/bladder and cerebral/mental FS. EDSS and FS scores are based on neurological examination for assessing its impairment in MS. Among eight FS, seven are ordinal clinical rating scales ranging from 0-5 or 6 with higher scale indicates overall functional impairment assessing Visual,Brain Stem,Pyramidal,Cerebellar,Sensory, Bowel/Bladder and Cerebral functions. Rating individual FS scores is used to rate EDSS in conjunction with observations and information concerning gait and use of assistance. EDSS is ordinal clinical rating scale ranging from 0 (normal neurological examination) to 10(death due to MS).
Time Frame: From randomization to end of study (Week 108)
Population: Full analysis set (FAS) included all participants randomized in the study.
Measure: Mean (99% Confidence Interval); unit: relapses per year
Arm/Group | Ponesimod 20 mg | Teriflunomide 14 mg
Number analyzed (Participants) | 567 | 566
relapses per year | 0.202 [0.165 to 0.246] | 0.290 [0.244 to 0.345]
Statistical Analysis 1: Comparison: Ponesimod 20 mg vs Teriflunomide 14 mg; Test type: Superiority; p = 0.0003, Negative binomial regression model; Rate ratio = 0.695, 99% CI 2-sided [0.536 to 0.902]

2. Secondary Outcome: Change From Baseline in Fatigue-related Symptoms as Measured by the Symptoms Domain of the Fatigue Symptom and Impact Questionnaire-Relapsing Multiple Sclerosis (FSIQ-RMS) Score to Week 108
Description: The FSIQ-RMS is a 20-item Patient Reported Outcomes (PRO) measure to evaluate fatigue-related symptoms and the impacts of those symptoms on the lives of people. The FSIQ-RMS symptom domain (FSIQ-RMS-S) consists of seven items assessing fatigue-related symptoms daily with a recall period of 24 hours measured on an 11-point numeric rating scale; the (normalized) symptom domain score ranges from 0 to 100 with a higher score indicating greater fatigue. This domain was completed on 7 consecutive days. A negative change from baseline indicates an improvement in fatigue symptoms.
Time Frame: Baseline to Week 108
Population: FAS included all participants randomized in the study. Here 'N' (number of participants analyzed) included all participants who were evaluable for this outcome measure with available baseline and at least one post-baseline assessment.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on scale
Arm/Group | Ponesimod 20 mg | Teriflunomide 14 mg
Number analyzed (Participants) | 449 | 458
score on scale | -0.01 [-1.60 to 1.58] | 3.56 [1.96 to 5.16]
Statistical Analysis 1: Comparison: Ponesimod 20 mg vs Teriflunomide 14 mg; Test type: Superiority; p = 0.0019, Mixed Models Analysis; Mean Difference (Final Values) = -3.57, 95% CI 2-sided [-5.83 to -1.32]

3. Secondary Outcome: Cumulative Number of Combined Unique Active Lesions (CUAL) Per Year From Baseline to Week 108
Description: CUALs was calculated as sum of new Gadolinium-enhanced (Gd+) T1 lesions plus new or enlarging T2 lesions (without double-counting of lesions) from baseline based on the Magnetic resonance imaging (MRI) scans up to Week 108. Average number of lesions per year were reported.
Time Frame: Baseline to Week 108
Population: FAS included all participants randomized in the study. Here 'N' (number of participants analyzed) signifies number of participants evaluable for this outcome measure.
Measure: Mean (95% Confidence Interval); unit: lesions per year
Arm/Group | Ponesimod 20 mg | Teriflunomide 14 mg
Number analyzed (Participants) | 539 | 536
lesions per year | 1.405 [1.215 to 1.624] | 3.164 [2.757 to 3.631]
Statistical Analysis 1: Comparison: Ponesimod 20 mg vs Teriflunomide 14 mg; Test type: Superiority; p < .0001, Negative binomial regression model; Rate Ratio = 0.444, 95% CI 2-sided [0.364 to 0.542]

4. Secondary Outcome: 12-Week Confirmed Disability Accumulation (CDA) Assessed From Baseline to EOS
Description: A 12-week CDA was defined as an increase of at least 1.5 in Expanded Disability Status Scale (EDSS) for participants with a baseline EDSS score of 0.0 or an increase of at least 1.0 in EDSS for participants with a baseline EDSS score of 1.0 to 5.0, or an increase of at least 0.5 in EDSS for participants with a baseline EDSS score greater than or equal to (>=) 5.5, which was confirmed after 12 weeks. Baseline EDSS was defined as the last EDSS score recorded prior to randomization. EDSS is an ordinal clinical rating scale ranging from 0 (normal neurological examination) to 10 (death due to MS).
Time Frame: Baseline to Week 60 and 108 Weeks
Population: FAS included all participants randomized in this study.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Ponesimod 20 mg | Teriflunomide 14 mg
Number analyzed (Participants) | 567 | 566
Percentage of Participants
  60 Weeks- from Kaplan Meier estimates | 7.6 [5.7 to 10.2] | 8.3 [6.3 to 11.0]
  108 Weeks- from Kaplan Meier estimates | 10.8 [8.4 to 13.7] | 13.2 [10.6 to 16.3]
Statistical Analysis 1: Comparison: Ponesimod 20 mg vs Teriflunomide 14 mg; Test type: Superiority; p = 0.2939, Log Rank; Hazard Ratio (HR) = 0.83, 95% CI 2-sided [0.58 to 1.18]

5. Secondary Outcome: 24-Week Confirmed Disability Accumulation (CDA) Assessed From Baseline to EOS
Description: A 24-week CDA was defined as an increase of at least 1.5 in EDSS for participants with a baseline EDSS score of 0.0 or an increase of at least 1.0 in EDSS for participants with a baseline EDSS score of 1.0 to 5.0, or an increase of at least 0.5 in EDSS for participants with a baseline EDSS score >= 5.5, which was confirmed after 24 weeks. Baseline EDSS was defined as the last EDSS score recorded prior to randomization. The EDSS is an ordinal scale ranging from 0 (normal neurological exam) to 10 (death to MS).
Time Frame: Baseline to 60 Weeks and 108 Weeks
Population: FAS included all participants randomized in this study.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Ponesimod 20 mg | Teriflunomide 14 mg
Number analyzed (Participants) | 567 | 566
Percentage of Participants
  60 Weeks- from Kaplan Meier estimates | 6.3 [4.6 to 8.7] | 6.9 [5.0 to 9.3]
  108 Weeks- from Kaplan Meier estimates | 8.7 [6.6 to 11.4] | 10.5 [8.2 to 13.4]
Statistical Analysis 1: Comparison: Ponesimod 20 mg vs Teriflunomide 14 mg; Test type: Superiority; p = 0.3720, Log Rank; Hazard Ratio (HR) = 0.84, 95% CI 2-sided [0.57 to 1.24]

ADVERSE EVENTS:
Time Frame: Up to 111 Weeks (From treatment start [Day 1] to end of treatment [Week 108] plus 15 days)
Description: Safety analysis set included all participants who received at least one dose of study treatment.
Arm/Group | Ponesimod 20 mg | Teriflunomide 14 mg
All-Cause Mortality (participants affected / at risk) | 0/565 | 2/566
Serious Adverse Events (participants affected / at risk) | 49/565 | 46/566
Other Adverse Events (participants affected / at risk) | 434/565 | 422/566
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ponesimod 20 mg (N=565) | Teriflunomide 14 mg (N=566)
Lymphadenitis (Blood and lymphatic system disorders) | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Atrial Fibrillation (Cardiac disorders) | 0 | 1
Coronary Artery Insufficiency (Cardiac disorders) | 0 | 1
Abdominal Pain (Gastrointestinal disorders) | 3 | 0
Bowel Movement Irregularity (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 0
Duodenal Ulcer Haemorrhage (Gastrointestinal disorders) | 0 | 1
Duodenitis (Gastrointestinal disorders) | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 1
Haemorrhoidal Haemorrhage (Gastrointestinal disorders) | 1 | 0
Intestinal Haemorrhage (Gastrointestinal disorders) | 1 | 0
Pancreatitis Acute (Gastrointestinal disorders) | 1 | 0
Biliary Colic (Hepatobiliary disorders) | 0 | 1
Cholecystitis Acute (Hepatobiliary disorders) | 0 | 1
Cholecystitis Chronic (Hepatobiliary disorders) | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 1 | 3
Drug-Induced Liver Injury (Hepatobiliary disorders) | 1 | 0
Hepatitis (Hepatobiliary disorders) | 0 | 1
Hepatitis Toxic (Hepatobiliary disorders) | 0 | 1
Abdominal Infection (Infections and infestations) | 1 | 0
Appendicitis (Infections and infestations) | 3 | 0
Bronchitis (Infections and infestations) | 0 | 1
Herpes Zoster (Infections and infestations) | 1 | 0
Lymph Node Abscess (Infections and infestations) | 0 | 1
Meningitis (Infections and infestations) | 0 | 1
Meningitis Enteroviral (Infections and infestations) | 0 | 1
Pilonidal Cyst (Infections and infestations) | 1 | 0
Salpingitis (Infections and infestations) | 0 | 1
Urinary Tract Infection (Infections and infestations) | 1 | 0
Vestibular Neuronitis (Infections and infestations) | 0 | 1
Concussion (Injury, poisoning and procedural complications) | 0 | 2
Fall (Injury, poisoning and procedural complications) | 0 | 1
Femur Fracture (Injury, poisoning and procedural complications) | 0 | 1
Fibula Fracture (Injury, poisoning and procedural complications) | 0 | 1
Jaw Fracture (Injury, poisoning and procedural complications) | 1 | 0
Ligament Injury (Injury, poisoning and procedural complications) | 1 | 0
Meniscus Injury (Injury, poisoning and procedural complications) | 0 | 1
Multiple Injuries (Injury, poisoning and procedural complications) | 1 | 0
Post Procedural Haematoma (Injury, poisoning and procedural complications) | 1 | 0
Soft Tissue Injury (Injury, poisoning and procedural complications) | 0 | 1
Toxicity to Various Agents (Injury, poisoning and procedural complications) | 0 | 1
Alanine Aminotransferase Increased (Investigations) | 0 | 2
Aspartate Aminotransferase Increased (Investigations) | 0 | 1
Hepatic Enzyme Increased (Investigations) | 1 | 0
Transaminases Increased (Investigations) | 0 | 1
Weight Decreased (Investigations) | 1 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Intervertebral Disc Protrusion (Musculoskeletal and connective tissue disorders) | 1 | 1
Myofascial Pain Syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Rheumatoid Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Spinal Pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Synovitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Eyelid Haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Invasive Ductal Breast Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Malignant Melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Pituitary Tumour Benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Squamous Cell Carcinoma of the Cervix (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Uterine Leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Clonic Convulsion (Nervous system disorders) | 1 | 0
Epilepsy (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 1 | 0
Ischaemic Stroke (Nervous system disorders) | 0 | 1
Loss of Consciousness (Nervous system disorders) | 0 | 1
Lumbar Radiculopathy (Nervous system disorders) | 2 | 1
Multiple Sclerosis (Nervous system disorders) | 0 | 1
Multiple Sclerosis Relapse (Nervous system disorders) | 1 | 1
Partial Seizures with Secondary Generalisation (Nervous system disorders) | 1 | 0
Restless Legs Syndrome (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 0
Trigeminal Neuralgia (Nervous system disorders) | 0 | 1
Conversion Disorder (Psychiatric disorders) | 0 | 1
Depression (Psychiatric disorders) | 0 | 1
Panic Attack (Psychiatric disorders) | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0
Proteinuria (Renal and urinary disorders) | 1 | 0
Renal Colic (Renal and urinary disorders) | 1 | 0
Tubulointerstitial Nephritis (Renal and urinary disorders) | 1 | 0
Ureterolithiasis (Renal and urinary disorders) | 0 | 1
Breast Cyst (Reproductive system and breast disorders) | 0 | 1
Endometrial Hyperplasia (Reproductive system and breast disorders) | 1 | 1
Endometriosis (Reproductive system and breast disorders) | 1 | 1
Menorrhagia (Reproductive system and breast disorders) | 1 | 0
Metrorrhagia (Reproductive system and breast disorders) | 0 | 2
Ovarian Cyst (Reproductive system and breast disorders) | 0 | 1
Pelvic Adhesions (Reproductive system and breast disorders) | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Abortion Induced (Surgical and medical procedures) | 2 | 0
Haemorrhoid Operation (Surgical and medical procedures) | 1 | 0
Hysterectomy (Surgical and medical procedures) | 1 | 0
Ligament Operation (Surgical and medical procedures) | 1 | 0
Uterine Dilation and Curettage (Surgical and medical procedures) | 0 | 1
Deep Vein Thrombosis (Vascular disorders) | 1 | 0
Hypertensive Crisis (Vascular disorders) | 1 | 1
Raynaud's Phenomenon (Vascular disorders) | 0 | 1
Thrombophlebitis Superficial (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ponesimod 20 mg (N=565) | Teriflunomide 14 mg (N=566)
Neutropenia (Blood and lymphatic system disorders) | 6 | 13
Vertigo (Ear and labyrinth disorders) | 13 | 7
Abdominal Pain (Gastrointestinal disorders) | 9 | 18
Abdominal Pain Upper (Gastrointestinal disorders) | 19 | 24
Constipation (Gastrointestinal disorders) | 16 | 21
Diarrhoea (Gastrointestinal disorders) | 20 | 44
Dyspepsia (Gastrointestinal disorders) | 13 | 13
Nausea (Gastrointestinal disorders) | 43 | 47
Vomiting (Gastrointestinal disorders) | 11 | 18
Asthenia (General disorders) | 11 | 18
Fatigue (General disorders) | 34 | 37
Pyrexia (General disorders) | 12 | 7
Bronchitis (Infections and infestations) | 26 | 24
Gastroenteritis (Infections and infestations) | 12 | 18
Influenza (Infections and infestations) | 24 | 23
Nasopharyngitis (Infections and infestations) | 109 | 95
Oral Herpes (Infections and infestations) | 17 | 21
Pharyngitis (Infections and infestations) | 14 | 14
Respiratory Tract Infection (Infections and infestations) | 17 | 16
Respiratory Tract Infection Viral (Infections and infestations) | 18 | 10
Rhinitis (Infections and infestations) | 12 | 17
Sinusitis (Infections and infestations) | 8 | 16
Tonsillitis (Infections and infestations) | 8 | 14
Upper Respiratory Tract Infection (Infections and infestations) | 60 | 59
Urinary Tract Infection (Infections and infestations) | 31 | 29
Alanine Aminotransferase Increased (Investigations) | 110 | 51
Aspartate Aminotransferase Increased (Investigations) | 36 | 19
C-Reactive Protein Increased (Investigations) | 12 | 7
Hepatic Enzyme Increased (Investigations) | 13 | 8
Weight Decreased (Investigations) | 6 | 14
Hypercholesterolaemia (Metabolism and nutrition disorders) | 13 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 17 | 15
Back Pain (Musculoskeletal and connective tissue disorders) | 33 | 38
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 20 | 17
Dizziness (Nervous system disorders) | 28 | 15
Headache (Nervous system disorders) | 64 | 72
Hypoaesthesia (Nervous system disorders) | 14 | 14
Paraesthesia (Nervous system disorders) | 17 | 28
Somnolence (Nervous system disorders) | 18 | 9
Anxiety (Psychiatric disorders) | 18 | 16
Depression (Psychiatric disorders) | 21 | 28
Insomnia (Psychiatric disorders) | 11 | 16
Cough (Respiratory, thoracic and mediastinal disorders) | 20 | 14
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 30 | 7
Alopecia (Skin and subcutaneous tissue disorders) | 18 | 72
Rash (Skin and subcutaneous tissue disorders) | 8 | 14
Hypertension (Vascular disorders) | 45 | 44

LIMITATIONS AND CAVEATS:
Low probability of this study to provide robust evaluation of ponesimod effect on disability accumulation compared to active comparator; study was not powered for this secondary endpoint. Impact of accelerated elimination procedure during safety follow-up: Accelerated elimination procedure for teriflunomide with cholestyramine/activated charcoal was frequently associated with benign, transient elevation in liver enzymes. Confounding effect of this procedure on assessing liver test was included.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested by the sponsor in writing, the investigator will withhold such publication for up to an additional 60 days.

DOCUMENTS (2):
  • Study Protocol (2018-12-05): https://cdn.clinicaltrials.gov/large-docs/44/NCT02425644/Prot_000.pdf
  • Statistical Analysis Plan (2019-06-20): https://cdn.clinicaltrials.gov/large-docs/44/NCT02425644/SAP_001.pdf